CLINICAL TRIAL: NCT01072344
Title: Long-Term Chamomile Therapy for Generalized Anxiety Disorder (GAD)
Brief Title: Long Term Chamomile Therapy for Anxiety
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AT005074
Record Dates: First submitted 2010-02-18; First posted 2010-02-22 (Estimated); Results first posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: Generalized Anxiety Disorder
Keywords: Anxiety; Chamomile; Herbal Remedy; Complementary and Alternative Medicine
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — Chamomile extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chamomile Extract (Experimental): Pharmaceutical grade oral chamomile extract.
  Interventions: Drug: Chamomile (Matricaria recutita)
- Placebo (Placebo Comparator): Pharmaceutical grade lactose monohydrate.
  Interventions: Drug: Chamomile (Matricaria recutita)

INTERVENTIONS:
Drug: Chamomile (Matricaria recutita) — 500 mg 3 times daily
  Other Names: Chamomile

SUMMARY:
Prior research has shown that chamomile may be an effective, short-term anti-anxiety treatment. This study will examine the initial and long-term benefits of chamomile extract therapy for the prevention of recurrent anxiety disorder.

DETAILED DESCRIPTION:
Anxiety disorders are among the most common psychiatric conditions. They affect up to 25% of the US adult population. Generalized anxiety disorder (GAD) is a chronic, recurrent form of the disorder. Although benzodiazepines and serotonin reuptake inhibitors have become the mainstay therapy of GAD, these drugs are often associated with unwanted side effects, habituation, and withdrawal symptoms. Many individuals decline using conventional drug therapy for financial, cultural, or personal reasons such as the stigma of mental illness. As a result, many individuals will seek alternative therapy for their anxiety symptoms. The identification of effective alternative therapies for GAD would be of particular relevance. Among alternative therapies for anxiety, chamomile has been used as a traditional herbal medicine for its calming effect. It is well tolerated and demonstrates pharmacological activity in animal models of anxiety. Despite its widespread use and availability, there has been only one clinical trial of chamomile safety and efficacy in GAD. The current application seeks to build upon the results of that prior chamomile study. In that 8-week, double-blind, placebo-controlled trial, we found a significant superiority of chamomile (vs. placebo) in reducing GAD symptoms. We also found chamomile to be exceedingly well tolerated (vs. placebo). The current application seeks to extend these promising preliminary results by conducting a randomized, double-blind, parallel group, placebo-substitution, long-term safety and efficacy study of chamomile in preventing GAD relapse. For specific aim #1 we will ask: "Does long-term chamomile therapy (vs. placebo) prolong the time to relapse of anxiety symptoms following recovery from GAD?" To answer this question, 180 patients with moderate to severe GAD will receive open-label chamomile extract 500-1,500 mg daily for 8 weeks. Responders to chamomile, who remain well for 4 additional weeks of consolidation therapy, will be randomized to double-blind continuation therapy with chamomile 500-1,500 mg daily or placebo for an additional 26 weeks. We hypothesize that continuation chamomile therapy will result in a prolonged time to relapse (vs. placebo). For specific aim #2 we will ask: "What is the relative safety and tolerability of long-term chamomile therapy (vs. placebo) in patients who have recovered from GAD?" To answer this question, we will examine the following outcome measures: (i) the proportion of patients in each treatment condition who relapse; (ii) the frequency, severity, and duration of treatment-emergent adverse events; (iii) the frequency of discontinuation symptoms during initial double-blind therapy; and, (iv) the frequency of early study discontinuation. We hypothesize that chamomile therapy will result in a lower proportion of anxiety relapses and a lower study discontinuation rate (vs. placebo). We further hypothesize that chamomile therapy will result in a similar frequency of discontinuation symptoms and treatment-emergent adverse events (vs. placebo).

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 18 years old (all races and ethnicity)
* DSM IV diagnosis of GAD as the primary anxiety disorder
* Baseline GAD-7 score ≥ 10
* Baseline CGI/S score at least 4
* Not taking anti-anxiety medication (e.g., Benzodiazepines, buspirone, antidepressants)
* Not taking antidepressant, mood stabilizer, or tranquilizer therapy for a prior DSM IV Axis I mood disorder that is in remission
* Able to understand and provide informed consent
* Able to participate in a 38-week study

Exclusion Criteria:

* Patients < 18 years old
* Primary DSM IV Axis I anxiety disorder other than GAD (e.g., panic disorder with or without agoraphobia, phobia disorder, acute stress disorder, social anxiety disorder, obsessive-compulsive disorder, post-traumatic stress disorder, substance-induced anxiety disorder)
* Current DSM IV Axis I psychotic disorder
* Substance abuse or dependence within the prior 3 months
* Current DSM IV Axis I bipolar or major depressive disorder [Note: Patients with co-morbid depressive disorder NOS (e.g., minor depression, recurrent brief depressive disorder, or premenstrual dysphoric disorder (PMDD)] will not be excluded
* Unstable medical condition
* Allergy to chamomile
* Documented allergy to plants of the asteraceae family (e.g., ragweed, asters, chrysanthemum)
* Allergic to mugwort or birch pollen
* Concurrent anti-anxiety tranquilizer, antidepressant or mood stabilizer therapy
* Concurrent use of over-the-counter anti-anxiety and/or antidepressant preparations (e.g., chamomile, St. John's Wort, kava kava)
* Concurrent use of established antidepressant, mood stabilizer, or tranquilizer therapy for pre-existing affective disorder. [Note: Patients with a history of affective disorder (in remission) who are not currently taking antidepressant, mood stabilizer, or tranquilizer therapy are not excluded from the trial]
* Women of child-bearing potential not willing to use a medically proven form of contraception
* Positive pregnancy test
* Actively suicidal or suicide attempt within the preceding 12 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun J Mao, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Depression Research Unit, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keefe JR, Guo W, Li QS, Amsterdam JD, Mao JJ. An exploratory study of salivary cortisol changes during chamomile extract therapy of moderate to severe generalized anxiety disorder. J Psychiatr Res. 2018 Jan;96:189-195. doi: 10.1016/j.jpsychires.2017.10.011. Epub 2017 Oct 16. PMID 29080520
- [Derived] Mao JJ, Xie SX, Keefe JR, Soeller I, Li QS, Amsterdam JD. Long-term chamomile (Matricaria chamomilla L.) treatment for generalized anxiety disorder: A randomized clinical trial. Phytomedicine. 2016 Dec 15;23(14):1735-1742. doi: 10.1016/j.phymed.2016.10.012. Epub 2016 Oct 24. PMID 27912875
- [Derived] Keefe JR, Amsterdam J, Li QS, Soeller I, DeRubeis R, Mao JJ. Specific expectancies are associated with symptomatic outcomes and side effect burden in a trial of chamomile extract for generalized anxiety disorder. J Psychiatr Res. 2017 Jan;84:90-97. doi: 10.1016/j.jpsychires.2016.09.029. Epub 2016 Sep 30. PMID 27716513
- See also: University of Pennsylvania Depression Research Unit Website — http://www.med.upenn.edu/dru

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study has 3 phases. The 1st phase is open label cham.(N=179), subjects meeting response criteria enter 2nd phase (N=93), the consolidation phase of open label chamomile. At the end of 2nd phase, if subjects still meet response criteria, they will enter the 3rd phase (N=93). In the 3rd phase, subjects will be randomized to chamomile vs. placebo.
Period: Overall Study
Arm/Group | Chamomile Extract | Placebo
Started | 46 | 47
Completed | 35 | 29
Not Completed | 11 | 18
Not completed — Relasped-reached end point | 7 | 12
Not completed — Protocol Violation | 1 | 2
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chamomile Extract | Placebo | Total
Number analyzed (Participants) | 46 | 47 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 42 | 82
  >=65 years | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (14.3) | 45.4 (16.1) | 47.3 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 31 | 65
  Male | 12 | 16 | 28
Region of Enrollment [Number; unit: participants]
  United States | 46 | 47 | 93

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse in Each Treatment Condition.
Description: The primary outcome was time to relapse during continuation therapy, analyzed using Cox proportional hazards. Relapse is dichotomously defined as an increase in CGI/S (a clinician-rated global measure of anxiety's severity) score from ≤ 3 (at study visit 6) to ≥ 4 (on two consecutive scheduled or unscheduled study visits ≥ 2 weeks apart) plus meeting DSM IV-TR criteria for GAD (minus the 6-month time criterion).
Time Frame: 26 weeks
Population: All 93 subjects started randomization phase of the study were included in the analysis
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Chamomile Extract | Placebo
Number analyzed (Participants) | 46 | 47
weeks | 11.4 (8.4) | 6.3 (3.9)

2. Secondary Outcome: The Proportion of Subjects in Each Treatment Condition Who Relapse.
Description: The proportion of subjects in each treatment condition who relapsed after randomization
Time Frame: 26 weeks
Population: During phase II consolidation phase, treatment responders were randomized to either 26 weeks of continuation chamomile therapy or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Chamomile Extract | Placebo
Number analyzed (Participants) | 46 | 47
Participants | 7 | 12

3. Secondary Outcome: Frequency, Severity, and Duration of Treatment-emergent Adverse Events.
Description: We will report the frequency, severity, and duration of treatment-emergent adverse events by treatment arm.
Time Frame: 26 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Chamomile Extract | Placebo
Number analyzed (Participants) | 46 | 47
Participants | 8 | 9

4. Secondary Outcome: Frequency of Discontinuation Symptoms at the Start of Double-blind Therapy in Each Treatment Condition.
Description: Discontinuation emergent signs and symptoms checklist (DESS) is a patient-rated measure of the presence and severity of discontinuation symptoms occurring after medication discontinuation. %
Time Frame: 26 weeks
Population: These are responders at the end of Phase II of the study and then were randomized in Phase III of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Chamomile Extract | Placebo
Number analyzed (Participants) | 46 | 47
Participants
  # of subject had no new symptoms after randomizat | 31 | 33
  # of subject had >=1 new symptom after randomizati | 14 | 11

5. Secondary Outcome: Frequency of Early Study Discontinuation in Each Treatment Condition.
Description: This is the # of subjects who discontinued the study during randomization phase due to other reasons.
Time Frame: 26 weeks
Population: These are responders at the end of Phase II of the study and were then randomized into Phase III of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Chamomile Extract | Placebo
Number analyzed (Participants) | 46 | 47
Participants
  # Lost to Follow-up | 3 | 4
  # withdrawn due to non-compliance | 1 | 2

ADVERSE EVENTS:
Arm/Group | Chamomile Extract | Placebo
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/47
Other Adverse Events (participants affected / at risk) | 8/46 | 9/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chamomile Extract (N=46) | Placebo (N=47)
taste perversion (Product Issues) | 1 (1) | 2 (2) — taste perversion caused by strong chamomile smell
Bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Decreased platelet count (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Drowsiness (Nervous system disorders) | 1 (1) | 0 (0)
Dry mouth (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Herbal taste (General disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ringing in ears (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Sleep paralysis (General disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No